CLINICAL TRIAL: NCT04639375
Title: A Proof-of-concept Study of Poliovirus Vaccine (IPV) Activity to Induce an Immune Response That Cross-reacts With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV-2)
Brief Title: Polio Vaccine (IPV) for SARS-CoV-2 and Prevention of Coronavirus Disease (COVID-19)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: E-MO Biology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EMO-001
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vaccinated with polio vaccine (IPV) (Experimental): All subjects will receive polio vaccine: IPV as manufactured by Sanofi Pasteur for distribution in the United States
  Interventions: Biological: Vaccinated with polio vaccine (IPV)

INTERVENTIONS:
Biological: Vaccinated with polio vaccine (IPV) — poliovirus vaccine (IPV) manufactured by Sanofi Pasteur for distribution in the United States

SUMMARY:
A total of 300 healthy volunteers between the ages of 18 and 80 with no previous history of COVID-19 will be entered into the study and will receive IPV by injection on Day 1. Blood specimens collected pre-inoculation will be tested for cross-reactivity to poliovirus and SARS-CoV-2 by Western blot. An additional specimen will be collected on Day 28 post-inoculation and, likewise tested for cross-reactivity to poliovirus and SARS-CoV-2.

The number of subjects with an immune response to SARS-CoV-2 antigens following inoculation with IPV will be summarized.

DETAILED DESCRIPTION:
A total of 300 healthy volunteers between the ages of 18 and 80 with no previous history of COVID-19 will be entered into the study and will receive IPV by injection on Day 1. Blood specimens collected pre-inoculation will be tested for cross-reactivity to poliovirus and SARS-CoV-2 by Western blot. An additional specimen will be collected on Day 28 post-inoculation and, likewise tested for cross-reactivity to poliovirus and SARS-CoV-2.

If the results from this study demonstrate that polio vaccine induces an immune response against both the immunogen (poliovirus) and SARS-CoV-2, the study may be amended after consultation with the Center for Biologics evaluation and research (CBER), to enroll an additional 275 subjects. Expansion of the original cohort will be stratified by age and race/ethnicity.

The number of subjects with an immune response to SARS-CoV-2 antigens following inoculation with IPV will be summarized.

Vaccination for poliomyelitis is part of routine childhood vaccination. Only IPV has been administered in the United States since the year 2000 as a series of 4 inoculations in childhood inducing an immunity which, although protective for years, wans over time and is, for the most part, undetectable in adults unless a booster is administered. United States residents are advised to receive a booster prior to travelling to countries where polio disease remains endemic.

Inactivated vaccines against RNA viruses (including Poliovirus and coronavirus) induce an immune response that recognizes the non-structural antigens of the inactivated viral particle. There is extensive homology between Poliovirus and SARS-CoV-2 RNA-dependent-RNA-polymerase (RdRp) both within the coding regions and illustrated in the 3-dimensional modeling. The homology between the viral epitopes may be sufficient such that adults who receive a polio booster develop an immune response that cross-reacts with SARS-CoV-2. Consequently, the neutralizing activity of antibodies raised to SARS-CoV-2 RdRp will be evaluated.To evaluate and characterize the immune response to SARS-CoV-2 elicited in adults by IPV.

Primary Objective: To evaluate whether an immune response to SARS-CoV-2 RdRp is induced in adults receiving a booster inoculation of IPV.

Secondary Objectives:: To evaluate the neutralizing activity of antibodies raised to SARS-CoV-2 RdRp

This is a single-site study in a clinic in San Diego California that routinely diagnoses and manages patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18-80
4. Female subjects of child-bearing potential must have a negative pregnancy test (point-of-care dipstick) prior to being vaccinated and be willing to use an effective method of birth control from the time of entry into the study and for 30 days following vaccination
5. In good general health with no active infectious disease as evidenced by medical history and directed physical examination.

Exclusion Criteria:

1. Known allergic reactions to components of the polio vaccine
2. Febrile illness within 14 days
3. Positive for SARS-CoV-2 antigenemia at any time prior to screening1
4. Positive for SARS-CoV-2 antibodies at any time prior to screening1
5. Subjects with fever > 101o F at screening
6. Subjects who respond yes to any of the following question:

   Have you experienced any of the following symptoms in the past 48 hours (14):
   * fever or chills
   * cough
   * shortness of breath or difficulty breathing
   * fatigue
   * muscle or body aches
   * headache
   * new loss of taste or smell
   * sore throat
   * congestion or runny nose
   * nausea or vomiting
   * diarrhea
7. Treatment with an investigational drug or other intervention within the 90 days prior to enrollment in this study
8. Inoculation with polio vaccine within the last 12 years
9. Women who are pregnant or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2022-06-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects with Antibodies to SARS-CoV-2 RdRp following IPV Vaccination | Day 28
  Percentage of all subjects vaccinated with IPV with antibodies to SARS-CoV-2 RdRp

SECONDARY OUTCOMES:
Determination of neutralizing titer of antibodies raised to SARS-CoV-2 following vaccination with polio vaccine | Day 28
  Antibodies raised following IPV vaccination will be evaluated for neutralizing titer to both polio virus and SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: John Andrews, Study Chair — E-MO Biology Inc
Locations (1):
- Rac Ii Md, National City, California, United States

IPD SHARING:
Plan to Share IPD: Undecided